CLINICAL TRIAL: NCT06748768
Title: The Effect of Omega 3 Supplements Comparison With Warm Compression in Patients With Dry Eye Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/043
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Chromosomes, Human, 1-3

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: group 1 — To determine the optimal treatment for dry eyes in term of cost effectiveness and time efficiency by comparing omega 3 supplements versus warm compression

SUMMARY:
dry eye disease is a common condition characterized by tear film instability and ocular surface inflammation. Omega 3 fatty acid and hot compression are two common tratement for dry eye diseases

DETAILED DESCRIPTION:
to investigate the cost effective and efficient treatment for dry eye diseases, During regular visit of patient assessment will be carried out to diagnose disease ,ocular findings and cause of visit .

ELIGIBILITY:
Inclusion Criteria:

* Young adults (20-39) years diagnosed with dry eyes and willingness to participate with no ocular surgery and infection from last 2 weeks Children

Exclusion Criteria:

* People having supplements
* Patients having diet with omega 3 for 1 month
* Patients who has undergone glaucoma treatment
* Already receiving treatment of dry eyes
* Patients with any ocular surgery

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: to check the he Effect of Omega 3 Supplements Comparison With Warm Compression in Patients With Dry Eye Disease
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
OSDI | 12 Months
  The OSDI score was grouped as per the following: normal (0-12 points), mild (13-22 points), moderate (23-32 points), and severe (33-100 points) [7]. Grouping for the number of years smoking was done in the following way: < 1 year, 1-5 years, 6-10 years, 11-15 years, 16-20 years, and 20+ years.

CONTACTS AND LOCATIONS:
Locations (1):
- Benazir Bhutu Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No